CLINICAL TRIAL: NCT02885857
Title: Safety and Efficacy of Shenyankangfu Tablets for Chronic Kidney Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chen Xiangmei (Other)
Collaborators: Tianjin TongRenTang Group Co., Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Chen Xiangmei, professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2015-023-02
Record Dates: First submitted 2015-06-03; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — shenyan kangfu

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Shenyan kangfu Tablets (Experimental): Shenyan Kangfu Tablets；Each weighing 0.48g；Oral；Once five, three times a day
  Interventions: Drug: Shenyan Kangfu Tablet

INTERVENTIONS:
Drug: Shenyan Kangfu Tablet — Observation period: 24 weeks. The dosage regimen: each piece weighs 0.48 g. 5 / time, 3 times daily, orally after dinner.

SUMMARY:
Safety and efficacy of long-term application of Shenyankangfu Tablets in Large sample of patients with chronic kidney disease.

DETAILED DESCRIPTION:
Research purpose: Safety and efficacy of long-term application of Shenyankangfu Tablets in Large sample of patients with chronic kidney disease.

The crowd: patients with primary glomerular nephritis, diabetic nephropathy patients.

Study design: a multicenter clinical study design, openness. The study drug: Shenyan Kangfu Tablets. Statistical analysis: Research plan is determined, by statistical professionals responsible for negotiation with the principal investigator for statistical analysis plan.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with primary glomerulonephritis or diabetic nephropathy;
2. Aged from 18 to 70 years，male or female
3. GFR≥45ml/min/1.73㎡
4. 0.5g≤24 hours proteinuria≤3.0g
5. glycated hemoglobin (HbAlc) ≤8% (This has been limited to patients with diabetic nephropathy)
6. Traditional Chinese medicine syndrome conform Qi-Yin Deficiency
7. Obtain the agreement of patients or their guardians, and signed informed consent file

Exclusion Criteria:

1. Secondary nephropathy
2. People allergic to Shenyankangfu tables
3. Combined with severe primary disease of heart, brain, liver and hematopoietic system, or other serious diseases can affect patient's life
4. Pregnant or lactating women
5. Be participating in another clinical study at the same period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
24-hour urinary protein excretion | Observation time: 24 weeks.Tested once every 12 weeks, it was detected three times

SECONDARY OUTCOMES:
Serum creatinine | Observation time: 24 weeks.Tested once every 12 weeks, it was detected three times
Glomerular filtration rate | Observation time: 24 weeks.Tested once every 12 weeks, it was detected three times
Albumin | Observation time: 24 weeks.Tested once every 12 weeks, it was detected three times
Glycated hemoglobin | Observation time: 24 weeks.Tested once every 24 weeks, were detected in 2 times
  Observations of the project value and the percentage change in value before and after the treatment.
Symptom scores | Observation time: 24 weeks.Tested once every 12 weeks, it was detected three times

OTHER OUTCOMES:
Routine blood test | Observation time: 24 weeks.Tested once every 12 weeks, it was detected three times
Routine urine test | Observation time: 24 weeks.Tested once every 12 weeks, it was detected three times
Liver function | Observation time: 24 weeks.Tested once every 12 weeks, it was detected three times
Renal function tests | Observation time: 24 weeks.Tested once every 12 weeks, it was detected three times
Potassium detection | Observation time: 24 weeks.Tested once every 12 weeks, it was detected three times
blood glucose testing | Observation time: 24 weeks.Tested once every 12 weeks, it was detected three times
Electrocardiograph | Observation time: 24 weeks.Tested once every 24 weeks, were detected in 2 times
chest radiography | Observation time: 24 weeks.Tested once every 24 weeks, were detected in 2 times
Adverse events / adverse reactions | Observation time: 24 weeks.Tested once every 24 weeks, were detected in 2 times
  Follow-up 3 times.Subject at any time to contact your doctor.

CONTACTS AND LOCATIONS:
Overall Officials: YongLi Zhan, investigator, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences; HongTao Yang, investigator, Principal Investigator — First Teaching Hospital of Tianjin University of Traditional Chinese Medicine; Meng Liang, investigator, Principal Investigator — 174th hospital of the People's Liberation Army; Lu Ma, investigator, Principal Investigator — Beidaihe Sanatorium of Beijing Military Mrca; LiQun Song, investigator, Principal Investigator — Heilongjiang University of Chinese Medicine; QiaoLing Zhou, investigator, Principal Investigator — Xiangya Hospital of Central South University; Ping Luo, investigator, Principal Investigator — Second Hospital of Jilin University; RongShan Li, investigator, Principal Investigator — Shanxi provincial peple's hospital; XiaoHong Cheng, investigator, Principal Investigator — Shaanxi Traditional Chinese Medicine Hospital; Jie Wu, investigator, Principal Investigator — Chinese PLA General Hospital
Locations (13):
- China (13):
  - National Clinical Research Center for Kidney Disease, State Key Laboratory of Kidney Disease, Department of Nephrology, Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Daping Hospital,Research Institute of Surgery Third Military Medical University, Chongqing, Chongqing Municipality
  - Fuzhou General Hospital Nanjing Military Command, Fuzhou, Fujian
  - 174th hospital of the People's Liberation Army, Xiamen, Fujian
  - Beidaihe Sanatorium of Beijing Military Mrca, Qinhuangdao, Hebei
  - Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang
  - Henan Provincial People'S Hospital, Zhengzhou, Henan
  - Shandong Province Hospital, Jinan, Shandong
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
  - LONGHUA Hospital Shanghai University of TCM, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - First Teaching Hospital of Tianjin University of TCM, Tianjin, Tianjin Municipality